CLINICAL TRIAL: NCT01931605
Title: Results of Selective Prostatic Arterial Embolization in Patients With Indwelling Urinary Catheter Due to Benign Prostatic Hyperplasia Refractory to Medical Treatment.
Acronym: Prost-EMBOL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Enrolling participants has halted prematurely and will not resume due to the Departure of the principal investigator
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012/173/HP
Record Dates: First submitted 2013-07-04; First posted 2013-08-29 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Embolization procedure (Experimental): selective prostatic arterial embolization using BeadBlock (Terumo) particules
  Interventions: Device: Prostatic arterial embolization using BeadBlock (Terumo)

INTERVENTIONS:
Device: Prostatic arterial embolization using BeadBlock (Terumo) — Selective Prostatic arterial embolization using BeadBlock (Terumo)particuls

SUMMARY:
Background: Patients with indwelling urinary catheter for chronic retention due to obstructive BPH refractory to medical therapy are candidates for prostatectomy still considered as the gold standard of treatment. Urinary tract infection, strictures, postoperative pain, incontinence, sexual dysfunction, anesthesiologist risk and blood loss are complications associated with surgery. Minimally invasive treatments were originally conceived as an attempt to offer equivalent efficacy without the burden and risk of operative morbidity. Recently, it was suggested that prostatic arterial embolization (PAE) to treat BPH might follow uterine artery embolization for uterine leiomyomas. Animal studies in pigs and dogs have shown that PAE is safe and can induce prostatic volume reduction. The first report of this technique in the management of BPH in humans was by DeMeritt et al, who reported a single case of BPH with obstructive symptoms and blood loss refractory to other treatments that was successfully managed by PAE with polyvinyl alcohol (PVA) particles.

Objective : We investigate whether PAE might be a feasible procedure as an alternative treatment option to treat urinary retention due to obstructive BPH. The primary objective is to evaluate the success rate of procedure defined when selective prostatic arterial catheterization and embolization were achieve and patients can be able to urinate after their urinary catheter has been removed.

Patients and methods : A monocentric prospective study is undertaken in 25 patients aged 50-85 years who present with indwelling urinary catheter due to obstructive BPH refractory to medical treatment with a clinical indication for surgery who agreed to undergo PAE. The study is approved by the hospital ethical committee and an informed consent form for PAE as an alternative treatment is signed by all participants.

Statistical analysis : The sample size has been calculated in order to have an estimated probability of success (corresponding of primary objective) of 50% (worst case) with 95% confidence intervals of 30 to 70. The two-sample t-test (and Wilcoxon rank-sum test) is used to compare the mean changes of the variables from baseline to 10, 30 and 90 days. Finally, the Chi-square test is used to test for adverse events at the end of follow-up. P ≤ 0.05 is indicative of statistically significant.

DETAILED DESCRIPTION:
Embolization is performed under local anesthesia in one day surgery unit by unilateral approach, usually the right femoral artery. Initially, pelvic angiography is performed to evaluate the iliac and prostatic arteries. Then, a 5-F catheter is introduced in right femoral artery to catheterize the left hypogastric artery and reach its anterior division. The inferior vesical artery and finally the prostatic vessels are selectively catheterized with a 3-F coaxial microcatheter. For embolization, nonspherical 100-300 μm PVA particles is used. The endpoint chosen for embolization is slow flow or near-stasis in the prostatic vessels with interruption of the arterial flow and prostatic gland opacification. When embolization of the left prostatic arteries was finished, the right prostatic arteries were embolized in the same way.

Urinary catheter is removed 10 days after the embolization procedure. Voiding trials is performed and the successfull urination after urethral catheter removal is defined as three consecutive spontaneous micturitions with postvoid residual less than 100% of each micturition volume. If the patient is unable to urinate, a urethral catheter will replace before hospitalization discharge and the patient will return to our outpatient clinic for another voiding trial until the end of protocol. Assessments were carried out 10, 30 and 90 days after initial embolization allocation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a urinary retention due to obstructive benign prostatic hyperplasia (BPH) confirmed by endoscopy,
* Patients aged 50-85 years,
* Patients with indwelling urinary catheter for at least 1 month,
* Patients with at least one failure of a trial without catheter despite alpha-blocker treatment for at least 72 hours,
* Patients informed about alternative treatment (transurethral resection of the prostate, laser prostatectomy, prostatic adenomectomy),
* Patients signed an informed consent form.

Exclusion Criteria:

* Prostate cancer (evaluated by PSA, physical examination, in all patients and by prostatic biopsy in suspicious cases).
* History of relevant neurological disease (e.g. multiple sclerosis, spinal cord injury, parkinson's disease).
* Patients who have on urodynamic investigation evidence of an atonic bladder.
* Urethral stricture
* Chronic persistent local pathology that may cause urinary symptoms (e.g. interstitial cystitis, tumor, bladder stone).
* Renal insufficiency stade 3 or 4 (creatinine clearance < 35 mL/min)
* Any allergy or contraindication to ciprofloxacin or drugs used in this protocole (xylocaine, Atarax, paracetamol, and nonsteroidal anti-inflammatory drug)
* Any allergy to intravenous contrast agent or iodine
* Thyrotoxicosis
* Concomitant use of tizanidine
* Patients participating to another research protocol

Ages: 50 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Procedural Success | Day 1
  * Procedural success was defined as cessation of extravasation and/or occlusion of the targeted vessel on postembolization arteriography.
  * Voiding diary : mictirution volume and postvoid residual volume measurements by ultrasonography

SECONDARY OUTCOMES:
success of the procedure : ability to urinate after their catheter | Day 10
  Ablation of Indwelling Urinary Catheter
success of the procedure : ability to urinate after their catheter | Day 90
  Ablation of Indwelling Urinary Catheter
success of the procedure : ability to urinate after their catheter | Day 30
  Ablation of Indwelling Urinary Catheter

CONTACTS AND LOCATIONS:
Overall Officials: Romain CAREMEL, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France